CLINICAL TRIAL: NCT05373901
Title: An Open-Label, Multi-Center, Single-Arm, Phase 1 Study Evaluating the Safety and Pharmacokinetics of Dinutuximab Beta as Maintenance Therapy in Chinese Patients With High-Risk Neuroblastoma
Brief Title: Evaluation of the Safety and Pharmacokinetics of Dinutuximab Beta As Maintenance Therapy in Chinese Participants With High-Risk Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-dinutuximab beta-101; CTR20221154 (Other: ChinaDrugTrials)
Record Dates: First submitted 2022-04-11; First posted 2022-05-13 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-06

CONDITIONS: High-risk Neuroblastoma
MeSH Terms: interventions — dinutuximab; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dinutuximab Beta + 13-cis-Retinoic Acid (Experimental): The study recruited participants who were hospitalized (with full resuscitation equipment) on Day 1 of each cycle and received continuous infusion of dinutuximab beta for 10 consecutive days in 35-day cycles. Participants could be discharged from the hospital at the investigator's discretion. Participants continued to receive 13-cis-retinoic acid orally for 14 days after completion of dinutuximab beta infusion (day 12-25 in each cycle).
  Interventions: Drug: Dinutuximab Beta; Drug: 13-cis-Retinoic Acid

INTERVENTIONS:
Drug: Dinutuximab Beta — Dinutuximab beta was administered intravenously at a dosage of 10 milligrams/ meters squared (mg/m2) per day for 10 consecutive days
Drug: 13-cis-Retinoic Acid — 13-cis-Retinoic Acid was administered orally at a daily total dose of 160 mg/m2, divided into approximately two equal doses given twice daily for 14 days following the conclusion of dinutuximab beta infusion.

SUMMARY:
This was an open-label, multi-center, single-arm, Phase 1 study. The purpose of this study was for evaluating the safety and pharmacokinetics of dinutuximab beta as maintenance therapy in Chinese participants with high-risk neuroblastoma

ELIGIBILITY:
1. Signed informed consent form (ICF) and ability to comply with study requirements
2. Age ≥ 12 months at consent
3. Diagnosis of high-risk neuroblastoma according to the International Neuroblastoma Staging System (INSS) criteria.
4. Participants who have previously received induction chemotherapy and achieved a partial or complete response followed by myeloablative therapy and stem cell transplantation. Stem cell transplantation should be completed within 120 days of dinutuximab beta first administration

Exclusion Criteria:

1. Hypersensitivity to ≥ 1 component of dinutuximab beta antibody or against mouse proteins
2. Actively progressive disease (not stabilized) or recurrent disease at the time of inclusion into the study
3. Previous treatment with anti-GD2 antibody before enrolling in this study

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Xinhua Hospital Affiliated To Shanghai Jiao Tong University School Of Medicine, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in three study centers across China. The study was conducted from June 7th, 2022, and completed on June 29, 2023.
Groups:
- Dinutuximab Beta + 13-cis-Retinoic Acid: The study recruited participants who were hospitalized (with full resuscitation equipment) on Day 1 of each cycle and received continuous infusion of dinutuximab beta for 10 consecutive days in 35-day cycles. Participants could be discharged from the hospital at the investigator's discretion. Participants continued to receive 13-cis-retinoic acid orally for 14 days after completion of dinutuximab beta infusion (day 12-25 in each cycle).
  Dinutuximab Beta: Dinutuximab beta was administered intravenously at a dosage of 10 milligrams/ meters squared (mg/m2/day) for 10 consecutive days.
  13-cis-Retinoic Acid: 13-cis-Retinoic Acid was administered orally at a daily total dose of 160 mg/m2, divided into approximately two equal doses given twice daily for 14 days following the conclusion of dinutuximab beta infusion.
Period: Overall Study
Arm/Group | Dinutuximab Beta + 13-cis-Retinoic Acid
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Dinutuximab Beta + 13-cis-Retinoic Acid: The study recruited participants who were hospitalized (with full resuscitation equipment) on Day 1 of each cycle and received continuous infusion of dinutuximab beta for 10 consecutive days in 35-day cycles. Participants could be discharged from the hospital at the investigator's discretion. Participants continued to receive 13-cis-retinoic acid orally for 14 days after completion of dinutuximab beta infusion (day 12-25 in each cycle).
  Dinutuximab Beta: Dinutuximab beta was administered intravenously at a dosage of 10 milligrams/ meters squared (mg/m2/day) for 10 consecutive days
  13-cis-Retinoic Acid: 13-cis-Retinoic Acid was administered orally at a daily total dose of 160 mg/m2, divided into approximately two equal doses given twice daily for 14 days following the conclusion of dinutuximab beta infusion.
Arm/Group | Dinutuximab Beta + 13-cis-Retinoic Acid
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.0 (1.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious treatment-emergent adverse event, characterized by type, frequency, severity (as graded by the National Cancer Institute- Common Terminology Criteria for Adverse Events Version 5.0 [NCI-CTCAE v 5.0]), timing, seriousness, relationship to study treatment, and other safety assessments.
Time Frame: From the first dose of study drug(s) to 40 days after the last dose; up to approximately 1 year and 1 month
Population: The Safety Analysis Set included all participants who received at least one dose of dinutuximab beta.
Measure: Count of Participants; unit: Participants
Arm/Group | Dinutuximab Beta + 13-cis-Retinoic Acid
Number analyzed (Participants) | 8
Participants
  Participants With At Least 1 TEAE | 8
  Participants with Serious TEAEs | 1

2. Primary Outcome: Area Under the Serum Concentration-time Curve From Zero to the Last Measurable Concentration (AUC0-t) of Dinutuximab Beta
Time Frame: From Cycle 1 Day 1 pre-dose to Cycle 2 Day 1 pre-dose (Each cycle is 35 Days)
Population: Pharmacokinetic (PK) Analysis Set was defined as participants who had at least 1 available postbaseline PK data in the Safety Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*micrograms/milliliter (h*ug/mL)
Arm/Group | Dinutuximab Beta + 13-cis-Retinoic Acid
Number analyzed (Participants) | 8
hours*micrograms/milliliter (h*ug/mL) | 3956.3 (33.11)

3. Primary Outcome: Area Under the Serum Concentration-time Curve From Zero to Infinity (AUC0-∞) of Dinutuximab Beta
Time Frame: From Cycle 1 Day 1 pre-dose to Cycle 2 Day 1 pre-dose (Each cycle is 35 Days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Dinutuximab Beta + 13-cis-Retinoic Acid
Number analyzed (Participants) | 8
h*ug/mL | 4228.6 (31.94)

4. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Dinutuximab Beta
Time Frame: From Cycle 1 Day 1 pre-dose to Cycle 2 Day 1 pre-dose (Each cycle is 35 Days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Dinutuximab Beta + 13-cis-Retinoic Acid
Number analyzed (Participants) | 8
ug/mL | 13.49 (32.682)

5. Primary Outcome: Time to Maximum Serum Concentration (Tmax) of Dinutuximab Beta
Time Frame: From Cycle 1 Day 1 pre-dose to Cycle 2 Day 1 pre-dose (Each cycle is 35 Days)
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Dinutuximab Beta + 13-cis-Retinoic Acid
Number analyzed (Participants) | 8
hours | 240.4 [168 to 252]

6. Primary Outcome: Half-Life (t1/2) of Dinutuximab Beta
Time Frame: From Cycle 1 Day 1 pre-dose to Cycle 2 Day 1 pre-dose (Each cycle is 35 Days)
Population: as for outcome 2
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Dinutuximab Beta + 13-cis-Retinoic Acid
Number analyzed (Participants) | 8
hours | 253.9 [200 to 332]

7. Primary Outcome: Clearance (CL) of Dinutuximab Beta
Time Frame: From Cycle 1 Day 1 pre-dose to Cycle 2 Day 1 pre-dose (Each cycle is 35 Days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Dinutuximab Beta + 13-cis-Retinoic Acid
Number analyzed (Participants) | 8
mL/h | 17.19 (34.627)

8. Primary Outcome: Volume of Distribution During Terminal Phase (Vz) of Dinutuximab Beta
Time Frame: From Cycle 1 Day 1 pre-dose to Cycle 2 Day 1 pre-dose (Each cycle is 35 Days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Dinutuximab Beta + 13-cis-Retinoic Acid
Number analyzed (Participants) | 8
mL | 6295.9 (48.87)

9. Primary Outcome: Volume of Distribution at Steady State (Vss) of Dinutuximab Beta
Time Frame: From Cycle 1 Day 1 pre-dose to Cycle 2 Day 1 pre-dose (Each cycle is 35 Days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Dinutuximab Beta + 13-cis-Retinoic Acid
Number analyzed (Participants) | 8
mL | 3594.0 (37.12)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events (AEs): From the first dose of study drug(s) to 40 days after the last dose; up to approximately 1 year and 1 month
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events include all randomized participants who received ≥ 1 dose of any study treatment AEs are defined as events that had an onset date or a worsening in severity from baseline (pretreatment) on or after the first dose of study treatment up to 40 days following study treatment discontinuation or initiation of a new anticancer therapy, whichever occurred first.
Groups:
- Dinutuximab Beta + 13-cis-Retinoic Acid: The study recruited participants who were hospitalized (with full resuscitation equipment) on Day 1 of each cycle and received continuous infusion of dinutuximab beta for 10 consecutive days in 35-day cycles. Participants could be discharged from the hospital at the investigator's discretion. Participants continued to receive 13-cis-retinoic acid orally for 14 days after completion of dinutuximab beta infusion (day 12-25 in each cycle).
  Dinutuximab beta was administered intravenously at a dosage of 10 mg/m2/day for 10 days
  13-cis-Retinoic Acid was administered orally at a daily total dose of 160 mg/m², divided into approximately two equal doses given twice daily for 14 days following the conclusion of dinutuximab beta infusion.
Arm/Group | Dinutuximab Beta + 13-cis-Retinoic Acid
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dinutuximab Beta + 13-cis-Retinoic Acid (N=8)
Pneumonia (Infections and infestations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dinutuximab Beta + 13-cis-Retinoic Acid (N=8)
Anaemia (Blood and lymphatic system disorders) | 5 (21)
Eosinophilia (Blood and lymphatic system disorders) | 2 (6)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 1 (2)
Dry eye (Eye disorders) | 2 (2)
Photophobia (Eye disorders) | 2 (2)
Swelling of eyelid (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (17)
Anal pruritus (Gastrointestinal disorders) | 1 (2)
Angular cheilitis (Gastrointestinal disorders) | 4 (12)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 6 (18)
Vomiting (Gastrointestinal disorders) | 4 (6)
Chills (General disorders) | 4 (8)
Face oedema (General disorders) | 2 (7)
Gait disturbance (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 8 (42)
COVID-19 (Infections and infestations) | 4 (8)
Catheter site infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Myringitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (8)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (14)
Alpha tumour necrosis factor increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (13)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood cholesterol increased (Investigations) | 1 (4)
Blood creatinine increased (Investigations) | 2 (2)
Blood fibrinogen decreased (Investigations) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 4 (10)
Brain natriuretic peptide increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 4 (10)
Electrocardiogram QT prolonged (Investigations) | 2 (3)
Fibrin D dimer increased (Investigations) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 5 (12)
Heart rate increased (Investigations) | 4 (55)
Interleukin level increased (Investigations) | 1 (1)
Interleukin-2 receptor increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (6)
Neutrophil percentage increased (Investigations) | 1 (2)
Oxygen saturation decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 4 (8)
Procalcitonin increased (Investigations) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (9)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 (13)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (11)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 1 (2)
Occipital neuralgia (Nervous system disorders) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (13)
Macule (Skin and subcutaneous tissue disorders) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 6 (12)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (4)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 (7)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 2 (4)
Haemorrhage (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 5 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights

DOCUMENTS (2):
  • Study Protocol (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT05373901/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT05373901/SAP_001.pdf